CLINICAL TRIAL: NCT05625568
Title: Phase 2, Double-Blind, Randomized, Placebo-Controlled Clinical Study of VYNT-0126 in the Treatment of Rett Syndrome in Adult Female Patients
Brief Title: Study of VYNT-0126 in the Treatment of Rett Syndrome in Adult Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vyant Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VYNT-0126-001
Record Dates: First submitted 2022-11-07; First posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 5 mg VYNT-0126 (Experimental)
  Interventions: Drug: VYNT-0126
- 10 mg VYNT-0126 (Experimental)
  Interventions: Drug: VYNT-0126

INTERVENTIONS:
Drug: VYNT-0126 — Liquid for oral administration once daily
  Arms: 10 mg VYNT-0126; 5 mg VYNT-0126
Drug: Placebo — Liquid for oral administration once daily
  Arms: Placebo

SUMMARY:
This is an exploratory, Phase 2, multicenter, double-blind, parallel-group, placebo-controlled study to assess the safety, tolerability, and efficacy of oral treatment with VYNT-0126 in female subjects 18-45 years of age with Rett syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Females age 18-45 (inclusive)
* Diagnosis of classic/typical Rett syndrome with a documented mutation of the MeCP2 gene
* Severity rating of between 10 and 36 (Rett Syndrome Natural History/Clinical Severity Scale)
* Concomitant medications (including approved medications for treatment of Rett syndrome) must be stable for >4 weeks prior to enrollment
* Able to receive liquid study drug orally or via gastrostomy tube (G-tube)

Exclusion Criteria:

* Actively undergoing neurological regression;
* Abnormal QT interval, prolongation or significant cardiovascular history
* Excluded concomitant medications
* Current clinically significant (as determined by the investigator). cardiovascular, endocrine, hepatic, renal, or respiratory disease
* Gastrointestinal disease which may interfere with the absorption, distribution, metabolism or excretion of the study medication
* History of, or current cerebrovascular disease or brain trauma
* History of, or current, malignancy
* Clinically significant abnormalities in safety laboratory tests, vital signs, or ECG, as measured at screening or baseline
* Any condition which in the investigator's opinion would affect the ability of the subject to participate in the study
* Allergy to VYNT-0126 or any ingredients of the liquid formulation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Through study completion, approximately 14 weeks
  Incidence of adverse events (AEs), including serious adverse events (SAEs), will be compared across the two VYNT-0126 doses and placebo. SAEs and AEs will be examined throughout the study.

SECONDARY OUTCOMES:
Change from Baseline in the Rett Syndrome Behavioral Questionnaire (RSBQ) | Obtained at baseline, end of dose titration, and end of treatment (approximately 14 weeks).
Change from Baseline in the 24-Item Motor-Behavioral Assessment (MBA) | Obtained at baseline, end of dose titration, and end of treatment (approximately 14 weeks).
Change from Baseline in Clinical Global Impression of Severity (CGI-S) | Obtained at baseline, end of dose titration, and end of treatment (approximately 14 weeks).
Clinical Global Impression of Improvement (CGI-I) | Obtained at the end of dose titration and end of treatment (approximately 14 weeks).

OTHER OUTCOMES:
Quantitative Electroencephalograms (EEGs) | Obtained at baseline, end of dose titration, and end of treatment (approximately 14 weeks).
  Quantitative EEGs will be explored as potential biomarkers of intervention effects on brain function and clinical severity.
Electrophysiological Evoked Potentials | Obtained at baseline, end of dose titration, and end of treatment (approximately 14 weeks).
  Evoked potential following auditory and visual stimuli will be explored as potential biomarkers of intervention effects on brain function and clinical severity.